CLINICAL TRIAL: NCT00585325
Title: Instilled Lidocaine vs Placebo for Pain Management During Vacuum Assisted Closure (VAC) Dressing Changes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-2004-0106
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instilled 1% Lidocaine (Experimental): 5 mg/kg of 1% lidocaine instilled into their VAC sponge ½ hour prior to VAC dressing change
  Interventions: Drug: Instilled 1% Lidocaine
- Instilled Placebo (0.9% Normal Saline) (Placebo Comparator): receive .9 normal saline instilled into their VAC sponge ½ hour prior to VAC dressing change
  Interventions: Other: Placebo (0.9% Normal Saline)

INTERVENTIONS:
Drug: Instilled 1% Lidocaine — 5 mg/kg of 1% lidocaine instilled into their VAC sponge ½ hour prior to VAC dressing change
  Other Names: Lidocaine
  Arms: Instilled 1% Lidocaine
Other: Placebo (0.9% Normal Saline) — .9 normal saline instilled into their VAC sponge ½ hour prior to VAC dressing change
  Other Names: Normal saline
  Arms: Instilled Placebo (0.9% Normal Saline)

SUMMARY:
Patients will be randomized prospectively to one of two groups. One group will receive 5 mg/kg of 1% lidocaine, and the other will receive .9 normal saline, instilled into their VAC sponge ½ hour prior to VAC dressing change. All patients will complete a pain assessment tool prior to receiving the instilled lidocaine/placebo, immediately after the procedure and 1 hour after the procedure. Pain scores will then be compared between the lidocaine and placebo groups.

Risks: Lidocaine toxicity is a potential risk, but 5 mg/kg of 1 % Lidocaine is below toxicity thresholds in an adult.

DETAILED DESCRIPTION:
• All Burn service patients (inpatients and outpatients in burn clinic) who are receiving VAC therapy will be screened for study inclusion criteria. Those with allergies to lidocaine will be excluded. Participants will be enrolled until a sample size of 80 wound VAC changes is achieved. Up to 4 VAC dressing changes can be included in this study per participant. Subjects will be randomized prospectively for each dressing change. Utilizing a randomized bracketed approach, patients will be assigned to one of two groups: Lidocaine group or Placebo group. The Pharmacy Research Center (PRC) will assign patient a study Identification (ID) number and record it along with their medical record number on the Master Study ID List. They will then randomize the participants by drawing randomly shuffled green vs white index cards. (40 white card = 0.9 normal saline and 40 green card = 5 mg/kg of 1% Lidocaine). They will draw up the appropriate amount of medication to be used, label it with the patients Medical Record (MR) #, date, and administration instructions and deliver it to the nurse who is doing the VAC dressing change. They will keep the Master Randomization Data Collection Tool in a locked drawer in her office.

ELIGIBILITY:
Inclusion Criteria:

* all burn service patients with a wound vac

Exclusion Criteria:

* allergy to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Schurr, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 patients were enrolled with 41 VAC dressing changes. Patients could be enrolled into more than one arm.
Units Other Than Participants: VAC dressing changes
Period: Overall Study
Arm/Group | Instilled 1% Lidocaine | Instilled Placebo (0.9% Normal Saline)
Started | 10; 20 VAC dressing changes | 13; 21 VAC dressing changes
Completed | 9; 14 VAC dressing changes | 12; 18 VAC dressing changes
Not Completed | 1; 6 VAC dressing changes | 1; 3 VAC dressing changes
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: VAC dressing changes
Groups:
- Total: Total of all reporting groups
Arm/Group | Instilled 1% Lidocaine | Instilled Placebo (0.9% Normal Saline) | Total
Number analyzed (Participants) | 9 | 12 | 21
Number analyzed (VAC dressing changes) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Pain During Dressing Change
Description: A pain assessment tool performed immediately after the dressing change was used to rate pain experienced during the dressing change. For this tool, pain was rated on a scale from 0-10 (0=no pain and 10=worst possible pain)
Time Frame: During dressing change
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: VAC dressing changes
Arm/Group | Instilled 1% Lidocaine | Instilled Placebo (0.9% Normal Saline)
Number analyzed (Participants) | 9 | 12
Number analyzed (VAC dressing changes) | 14 | 18
units on a scale | 6.36 (2.56) | 6.94 (3.11)

ADVERSE EVENTS:
Arm/Group | Instilled 1% Lidocaine | Instilled Placebo (0.9% Normal Saline)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes